CLINICAL TRIAL: NCT00829127
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Oral Doses of AZD8075 in Healthy Male Volunteers
Brief Title: AZD8075 Study to Assess the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Oral Doses of AZD8075 in Healthy Male Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to termination of study D3801C00001, due to reports of turbid urine.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D3801C00004; EudraCt No.2008-006550-17
Record Dates: First submitted 2009-01-20; First posted 2009-01-26 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD8075
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8075 — single dose, oral suspension, on Day 1. Repeated dosing will commence on Day 3 once daily for 14 days. The planned starting dose will be 35 mg with up to 2 dose escalations not exceeding AstraZeneca pre-defined upper exposure limits or the exposure obtained so far in the SAD study.
  Arms: 1
Drug: Placebo — Oral suspension
  Arms: 2

SUMMARY:
The aims of the study are to evaluate the safety, tolerability and pharmacokinetics of AZD8075 in healthy male subjects at increasing doses when given for 14 days

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures
* Have a body mass index (BMI) between 19 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg
* Be non-smoker or ex-smoker who has stopped smoking (or using other nicotine products) for >6 months prior to study start

Exclusion Criteria:

* Any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the result of the study, or the subject's ability to participate
* Any clinically relevant abnormal findings in phys.examination, clinical chemistry, haematology, urinalysis, vital signs or ECG at baseline, which, in the opinion of the investigator, may put the subject at risk because of his participation in the study
* Participation in another investigational drug study within 3 months before Visit 2 or participation in a method development study (no drug) 1 month prior to Visit 2

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Safety variables (ECG, adverse events, blood pressure, pulse, body temp, safety lab) | daily

SECONDARY OUTCOMES:
characterise the multiple dose PK of AZD8075 and assess the time required to reach steady state, the degree of accumulation and the time dependency of the PK | daily

CONTACTS AND LOCATIONS:
Overall Officials: Eva Pettersson, Study Director — AstraZeneca R&D, Lund, Sweden; Wolfgang Kühn, Principal Investigator — Quintiles, Uppsala, Sweden